CLINICAL TRIAL: NCT05639985
Title: The Prevalence of Malnutrition and Sarcopenia in Swiss Rehabilitation Settings
Acronym: Malnut-Reha
Status: Completed | Type: Observational
Sponsor: Undine Lehmann, Dr. (Other)
Collaborators: Berner Reha Zentrum AG (Other); Klinik Barmelweid (Other); University Department of Geriatric Medicine FELIX PLATTER (Other); Zürcher RehaZentrum Wald (Other); Rehab Basel (Other)
Responsible Party: Sponsor-Investigator, Undine Lehmann, Dr., Lecturer, Bern University of Applied Sciences
Organization: Bern University of Applied Sciences (Other)
Other Study IDs: 2022-01098
Record Dates: First submitted 2022-10-28; First posted 2022-12-07 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Malnutrition; Sarcopenia
Keywords: malnutrition; sarcopenia; rehabilitation; prevalence; Nutritional Risk Screening; handgrip strength
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to identify the prevalence of malnutrition and sarcopenia in patients admitted in Swiss rehabilitation centers. Furthermore, the aim is to investigate the changes of selected malnutrition and sarcopenia parameters over the length of the rehabilitation stay.

DETAILED DESCRIPTION:
The project aims to investigate the prevalence of malnutrition and sarcopenia in the rehabilitation setting. A cross-sectional national multicenter study will be conducted in five rehabilitation centers in Switzerland, including 80 - 130 participants per center for the primary objective (prevalence study). Patients will be screened for malnutrition and sarcopenia with established screening tools and if an elevated risk is observed, diagnosis will be confirmed and severity investigated according to international guidelines. Furthermore, the evolution of selected malnutrition and sarcopenia parameters over the rehabilitation stay should be assessed.

ELIGIBILITY:
Inclusion Criteria:

Patients treated in the following groups of rehabilitations will be included:

* Geriatric rehabilitation
* Pulmonal rehabilitation
* Cardiovascular rehabilitation
* Neurological rehabilitation
* Musculoskeletal rehabilitation
* Internistic rehabilitation and oncological rehabilitation

Exclusion criteria:

* Inability to give informed consent
* Inability to follow study procedures (e.g., due to delirium or language barriers)
* Expected life expectancy < 3 months and/or palliative care
* Isolation for example due to Covid-19 infection or tuberculosis
* Severe dehydration/ volume overload
* Medical conditions that prevent conducting a Bioelectrical Impedance Analysis (BIA) measurement (e.g. non-removable plasters or bandages at feet or hands) or defibrillator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inpatients in rehabilitation clinic
Sampling Method: Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of malnutrition - Risk for malnutrition | Within 7 days after admission
  The risk for malnutrition will be screened by the Nutritional Risk Screening (NRS-2002, in points). NRS has a scale from 0 to 7 points; higher points indicate a higher risk for malnutrition.
Body weight | Within 7 days after admission
  (in kg)
Height | Within 7 days after admission
  (in cm)
Body Mass Index | Within 7 days after admission
  (calculated by weight and height in kg/m2)
Weight loss | Within 7 days after admission
  Weight loss (in percent in six categories - <5 percent within the last 6 months, 5-10 percent within the last 6 months, >10 percent within the last 6 months; <10 percent in more than 6 months, 10 -20 percent in more than 6 months, >20 percent in more than 6 months)
Reduced energy intake | Within 7 days after admission
  Reduced energy intake (in percent of intake versus requirement in three categories: less than 50 percent of energy requirement covered for more than 1 week, any reduced energy intake versus requirement for >2 weeks, no reduced energy intake)
Muscle mass by Bioelectrical Impedance Analysis (BIA) - Part 1 | Within 7 days after admission
  Resistance (in Ohm) and Reactance (in Ohm)
Muscle mass by Bioelectrical Impedance Analysis (BIA) - Part 2 | Within 7 days after admission
  Resistance (in Ohm) and Reactance (in Ohm) measured with BIA are combined with further information on weight, height, sex and age to calculate the appendicular skeletal muscle mass index (in kg/m2)
Prevalence of malnutrition - Confirmed diagnosis and severity of malnutrition | Within 7 days after admission
  In case of positive screening, diagnosis of malnutrition will be confirmed and severity assessed according to the Global Leadership Initiative on Malnutrition (GLIM) criteria using the following measures described above: weight (in kg); height (in cm); Body Mass Index (calculated by weight and height in kg/m2); weight loss (in percent in six categories - <5 percent within the last 6 months, 5-10 percent within the last 6 months, >10 percent within the last 6 months; <10 percent in more than 6 months, 10 -20 percent in more than 6 months, >20 percent in more than 6 months); reduced energy intake (in percent of intake versus requirement in three categories: less than 50 percent of energy requirement covered for more than 1 week, any reduced energy intake versus requirement for >2 weeks, no reduced energy intake); Bioelectrical impedance analysis for muscle mass: resistance (in Ohm), reactance (in Ohm), Appendicular skeletal muscle mass index (in kg/m2)
Prevalence of malnutrition - overall | Calculated through study completion after five months recruitment duration
  Overall prevalence of malnutrition will be reported in percent

SECONDARY OUTCOMES:
Prevalence of sarcopenia - Risk for sarcopenia by SARC-F | Within 7 days after admission
  according to European Working Group on Sarcopenia in Older People (EWGSOP2) criteria. Screening will be performed by the Strength, assistance with walking, rising from a chair, climbing stairs, and falls (SARC-F) questionnaire (in points). SARC-F has a scale from 0 - 10 with higher score indicating higher risk for sarcopenia.
Prevalence of sarcopenia - Risk for sarcopenia by handgrip strength | Within 7 days after admission
  according to European Working Group on Sarcopenia in Older People (EWGSOP2) criteria. Screening will be performed by handgrip strength (in kPa)
Prevalence of sarcopenia - Risk for sarcopenia | Within 7 days after admission
  according to European Working Group on Sarcopenia in Older People (EWGSOP2) criteria. Screening will be performed by Chair Stand Test (in seconds)
Prevalence of sarcopenia - Diagnosis of sarcopenia | Within 7 days after admission
  In case of positive screening, muscle mass will be measured by BIA via resistance (in Ohm), reactance (in Ohm). Resistance (in Ohm) and Reactance (in Ohm) measured by BIA is combined with further information on weight, height, sex and age to calculate the appendicular skeletal muscle mass index in kg/m2. Diagnosis is confirmed if the appendicular skeletal muscle mass index is below a threshold (<7.0 kg/m2 for male and < 5.5. kg/m2 for female).
Prevalence of sarcopenia - Severity of sarcopenia | Within 7 days after admission
  In case of positive screening, severity of sarcopenia will be analysed by Timed Up and Go Test (in seconds).
Prevalence of sarcopenia - Overall | Calculated through study completion after five months recruitment duration
  Overall prevalence of sarcopenia will be reported in percent
Changes of handgrip strength between admission and discharge of rehabilitation | At admission and 21 days after admission (or, if admission occurs before 21 days and the length of stay was at least 14 days than within 3 days before discharge)
  Handgrip strength (in kPa)
Changes of body weight between admission and discharge of rehabilitation | At admission and 21 days after admission (or, if admission occurs before 21 days and the length of stay was at least 14 days than within 3 days before discharge)
  body weight (in kg)
Changes of BMI between admission and discharge of rehabilitation | At admission and 21 days after admission (or, if admission occurs before 21 days and the length of stay was at least 14 days than within 3 days before discharge)
  BMI (calculated in kg/m2)
Changes of Functional Independence Measure between admission and discharge of rehabilitation | At admission and 21 days after admission (or, if admission occurs before 21 days and the length of stay was at least 14 days than within 3 days before discharge)
  Functional Independence Measure (FIM) (in points). FIM has a scale from 18 to 126 points. Higher points indicate a higher independence for activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Thimo Marcin, Dr., Principal Investigator — Berner Reha Zentrum
Locations (5):
- Switzerland (5):
  - Klinik Barmelweid AG, Barmelweid
  - REHAB Basel, Basel
  - University Department of Geriatric Medicine FELIX PLATTER, Basel
  - Berner Reha Zentrum AG, Heiligenschwendi
  - Zürcher RehaZentren - Klinik Wald, Wald

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats A, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee; GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. Clin Nutr. 2019 Feb;38(1):1-9. doi: 10.1016/j.clnu.2018.08.002. Epub 2018 Sep 3. PMID 30181091
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673